CLINICAL TRIAL: NCT06055179
Title: Mechanistic and Pharmacokinetic Studies of Classical Chinese Formula Xiao Chai Hu Tang (XCHT) Against Irinotecan-Induced Gut Toxicities(Clinical Study Part:Randomized Controlled Trial)
Brief Title: XCHT for Irinotecan-Induced Gut Toxicities (Randomized Controlled Trial)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Guangzhou University of Traditional Chinese Medicine (Other)
Collaborators: University of Houston (Other)
Responsible Party: Principal Investigator, Haibo Zhang, Professor, Guangzhou University of Traditional Chinese Medicine
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2021KT1005-2; 81961128028 (Other Grant/Funding Number: National Nature Science Fundation of China)
Record Dates: First submitted 2023-09-09; First posted 2023-09-26 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2024-06

CONDITIONS: Xiao Chai Hu Tang; Irinotecan-induced Diarrhea
Keywords: Malignant tumor; Irinotecan-induced diarrhea; Xiao Chai Hu Tang; Classical Chinese Formula; pharmacokinetic mechanism
MeSH Terms: conditions — Neoplasms | interventions — shosaiko-to; Long-Term Synaptic Depression; Raloxifene Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Patients will be randomly assigned to XCHT/placebo groups, at a 1:1 ratio, using a central randomization system provided by the TCM clinical study methodology group of Guangdong Provincial Hospital of Chinese Medicine. This group is also responsible for blinding, including keeping the blinding codes, supervision, and quality control of blinding, by allocating drug codes for each patient. Investigators will dispense the drug according to the drug codes. The investigators, the study subjects, the care givers, and the outcome assessors will be blinded to the assigned group of subjects.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- XCHT group (Experimental): Patients will be administered with XCHT (9 g, qd, po) for 5 days each cycle of irinotecan chemotherapy for 3 cycles. The XCHT administration begins 3 days before chemotherapy in each cycle, that is the chemotherapy begins on the 4th day of XCHT administration. Plasma will be collected for pharmacokinetic testing (using raloxifene 60mg po as probe), on the day before chemotherapy, that is on the 3rd day of XCHT administration in each cycle.
  Interventions: Drug: Xiao Chai Hu Tang (XCHT); Drug: Irinotecan regimen; Other: Raloxifene
- Placebo group (Placebo Comparator): Patients will be administered with placebo (9 g, qd, po) for 5 days each cycle of irinotecan chemotherapy for 3 cycles. The placebo administration begins 3 days before chemotherapy in each cycle, that is the chemotherapy begins on the 4th day of placebo administration. Plasma will be collected for pharmacokinetic testing (using raloxifene 60mg po as probe), on the day before chemotherapy, that is on the 3rd day of placebo administration in each cycle.
  Interventions: Drug: Placebo; Drug: Irinotecan regimen; Other: Raloxifene

INTERVENTIONS:
Drug: Xiao Chai Hu Tang (XCHT) — XCHT 9g, po qd, 3 days before each cycle of chemotherapy for 5 days, for 3 cycles of chemotherapy.
  Other Names: Xiao Chai Hu Tang granules from Nin Jiom Medicine Manufactory (Hong Kong) Ltd
  Arms: XCHT group
Drug: Placebo — Placebo 9g, po qd, 3 days before each cycle of chemotherapy for 5 days, for 3 cycles of chemotherapy.
  Other Names: Placebo provided by Nin Jiom Medicine Manufactory (Hong Kong) Ltd
  Arms: Placebo group
Drug: Irinotecan regimen — Patients will receive 3 cycles of irinotecan chemotherapy. FOLFIRI regimen:irinotecan (180 mg/m2) intravenous (IV) for over 90 minutes on Day 1. Folinic acid (400 mg/m2) IV over 2 hours on Day 1. 5-fluorouracil (5-FU) IV bolus (400 mg/m2) over 5 minutes on Day 1, followed by 5-FU (2400 mg/m2) IV continuously for 46-48 hours. Every 2 weeks.
  mXELIRI regimen:irinotecan (200 mg/m2) intravenous (IV) for over 90 minutes on Day 1. Capecitabine (800 mg/m²) PO bid on day 1-14. Every 3 weeks.
  CapIRI regimen:irinotecan (180 mg/m2) intravenous (IV) for over 90 minutes on Day 1. Capecitabine (1000 mg/m²) PO bid on day 1-14. Every 3 weeks.
  FOLFOXIRI regimen:irinotecan (165 mg/m2) intravenous (IV) for over 90 minutes on Day 1. Oxaliplatin (85 mg/m2) intravenous (IV) for over 2 hours on Day 1.Folinic acid (400 mg/m2) IV over 2 hours on Day 1, followed by 5-FU (2400 - 3200 mg/m2) IV continuously for 48 hours. Every 2 weeks.
Other: Raloxifene — Raloxifene 60mg po, used as probe for pharmacokinetic testing, on Day 3 (the day before chemotherapy), for 3 cycles of chemotherapy.

SUMMARY:
Randomized double-blind placebo-controlled trial (RCT) study, to determine the impact of XCHT on irinotecan-induced severe delayed-onset diarrhea (SDOD), and to determine the feasibility of using plasma raloxifene-4'-glucuronide as a probe for intestinal UGT activity.

DETAILED DESCRIPTION:
A total of 98 patients, who are planning to recieve at least 3 cycles of irinotecan chemotherapy, will be randomly assigned, at a 1:1 ratio, to XCHT group or placebo group, using a central randomization system. Patients will be administered with XCHT/placebo (9 g, qd, po) for 5 days each cycle of chemotherapy for 3 cycles. The XCHT/placebo administration begins 3 days before chemotherapy in each cycle, that is the chemotherapy begins on the 4th day of XCHT/placebo administration. Plasma will be collected for pharmacokinetic testing (using raloxifene 60mg po as probe), on the day before chemotherapy, that is on the 3rd day of XCHT/placebo administration in each cycle. The purpose of this study includes 1) to determine the safety and efficacy of XCHT for prevention of irinotecan-induced diarrhea; 2) to determine the PK profile of SN-38, SN-38G, raloxifene, raloxifene-glucuronide, and XCHT components; and 3) to validate the use of raloxifene-4'G as a probe for irinotecan-induced diarrhea.

ELIGIBILITY:
Inclusion criteria:

1. Malignant tumor confirmed by histology or cytology;
2. Age ≥ 18 years old, ≤ 75 years old;
3. ECOG score of the patient ≤ 2 points;
4. Patients who have diarrhea worse than grade 2 due to irinotecan chemotherapy (the last dose of irinotecan is administered within 1 month);
5. Patients who plan to receive 3 cycles of irinotecan chemotherapy (the dose of irinotecan ≥ 125mg/m2);
6. Normal organ functions which can meet the requirements for systemic chemotherapy:

   * Normal bone marrow function: absolute neutrophil count (ANC) ≥ 1.5×109/L, PLT ≥ 100×109/L, hemoglobin ≥ 90g/L;
   * Normal renal functions: serum creatinine ≤ 1.5mg/dl (133μmol/L) and/or creatinine clearance ≥ 60ml/min;
   * Normal hepatic functions: total serum bilirubin level ≤ 1.5 times of the upper limit of normal value (ULN), serum aspartate aminotransferase (AST) & alanine aminotransferase (ALT) ≤ 2.5× ULN; AST & ALT ≤ 5 × ULN if abnormal hepatic functions are caused by a potentially malignant tumor.
7. Patients who can understand and complete the questionnaires in the case report form;
8. Patients who can understand and sign the informed consent form, is well compliant, and can be followed up.

Exclusion Criteria:

1. Patients with diagnosed depression, obsession or/and schizophrenia;
2. Patients with diagnosed inflammatory bowel diseases (including Crohn's disease, ulcerative colitis)
3. Patient with active tuberculosis and other uncontrolled infections;
4. Patient who has previously received radiotherapy on the abdominal cavity or pelvic cavity;
5. Pregnant or lactating women;
6. Patient who previously had or is now having thromboembolic events.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Estimated)
Dates: Start 2024-03-08 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of diarrhea (grade ≥2) | Through study completion, an average of 2 months
  The diarrhea severity will be evaluated following standard criteria in NCI-CTC AE 5.0 Grade 2 is defined as Stool is increased by 4-6 times each day relative to baseline; discharge from stoma moderately increased.

SECONDARY OUTCOMES:
Incidence of diarrhea (grade ≥3) | Through study completion, an average of 2 months
  The diarrhea severity will be evaluated following standard criteria in NCI-CTC AE 5.0
Incidence of other chemo-related adverse effects | Through study completion, an average of 2 months
  Other adverse reactions will be evaluated following standard criteria in NCI-CTC AE 5.0
Occult blood test for stool | Through study completion, an average of 2 months
  Occult blood test for stool, reported as negative, weak positive, and positive.
PK parameters(Cmax) | The blood samples (2.0 ml) will be collected at 4 points for each cycle(hour 0, hour 1, hour 2, hour 4 after raloxifene administration)
  Cmax ,if with complete data, in each cycle of Cmax for XCHT and their metabolites (14 compounds) and intestinal UGT enzyme probe (raloxifene and metabolites)
PK parameters(AUC) | The blood samples (2.0 ml) will be collected at 4 points for each cycle(hour 0, hour 1, hour 2, hour 4 after raloxifene administration)
  AUC 0-24hr, if with complete data, in each cycle of AUC0-24hr for XCHT and their metabolites (14 compounds) and intestinal UGT enzyme probe (raloxifene and metabolites)
PK parameters(T1/2) | The blood samples (2.0 ml) will be collected at 4 points for each cycle(hour 0, hour 1, hour 2, hour 4 after raloxifene administration)
  T1/2, if with complete data, in each cycle of T1/2 for XCHT and their metabolites (14 compounds) and intestinal UGT enzyme probe (raloxifene and metabolites)

CONTACTS AND LOCATIONS:
Overall Officials: Haibo Zhang, Prof., Principal Investigator — Guangdong Provincial Hospital of Traditional Chinese Medicine
Locations (1):
- Guangdong Provincial Hospital of Traditional Chinese Medicine, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No